CLINICAL TRIAL: NCT04817202
Title: hzVSF-v13 - A Phase I, Double-blind, Placebo-controlled, Single and Multiple Dose Study to Investigate Safety, Tolerability and Pharmacokinetics After Intravenous and Subcutaneous Administration in Healthy Adults
Brief Title: Safety, Tolerability, Pharmacokinetics of hzVSf-v13 in Healthy Adults (Intravenous and Subcutaneous Administration)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: hzVSF_v13-0002
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Injections, Subcutaneous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Group A1 (hzVSF-v13 50mg, intravenous, single dose) (Experimental): Single administration (intravenous) of 50mg hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13 (intravenous, single dose)
- Group A2 (hzVSF-v13 100mg, intravenous, single dose) (Experimental): Single administration (intravenous) of 100mg hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13 (intravenous, single dose)
- Group A3 (hzVSF-v13 200mg, intravenous, single dose) (Experimental): Single administration (intravenous) of 200mg hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13 (intravenous, single dose)
- Group A4 (hzVSF-v13 400mg, intravenous, single dose) (Experimental): Single administration (intravenous) of 400mg hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13 (intravenous, single dose)
- Group A5 (hzVSF-v13 800mg, intravenous, single dose) (Experimental): Single administration (intravenous) of 800mg hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13 (intravenous, single dose)
- Group A6 (hzVSF-v13 1200mg, intravenous, single dose) (Experimental): Single administration (intravenous) of 1200mg hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13 (intravenous, single dose)
- Group A7 (hzVSF-v13 100mg, subcutaneous, single dose) (Experimental): Single administration (subcutaneous) of 100mg hzVSF-v13 on Day 1.
  Interventions: Drug: hzVSF-v13 (subcutaneous, single dose)
- Group B1 (hzVSF-v13 100mg, intravenous, multiple dose) (Experimental): Multiple administration (intravenous) of 100mg hzVSF-v13 on Day 1, Day 15, Day 29, Day 43, Day 57.
  Interventions: Drug: hzVSF-v13 (intravenous, multiple dose)
- Group B2 (hzVSF-v13 400mg, intravenous, multiple dose) (Experimental): Multiple administration (intravenous) of 400mg hzVSF-v13 on Day 1, Day 15, Day 29, Day 43, Day 57.
  Interventions: Drug: hzVSF-v13 (intravenous, multiple dose)
- Placebo (intravenous, single dose) (Placebo Comparator): Single administration (intravenous) of placebo on Day 1.
  Interventions: Drug: Placebo (intravenous, single dose)
- Placebo (subcutaneous, single dose) (Placebo Comparator): Single administration (subcutaneous) of placebo on Day 1.
  Interventions: Drug: Placebo (subcutaneous, single dose)
- Placebo (intravenous, multiple dose) (Placebo Comparator): Multiple administration (intravenous) of placebo on Day 1, Day 15, Day 29, Day 43, Day 57.
  Interventions: Drug: Placebo (intravenous, multiple dose)

INTERVENTIONS:
Drug: hzVSF-v13 (intravenous, single dose) — Dosage form: 50mg / 100mg / 200mg / 400mg / 800mg /1200mg of hzVSF-v13 (40 mg/mL in a 5 mL vial) Route: Intravenous Frequency: Dose at Day 1 (single administration)
  Other Names: a humanized monoclonal antibody (mAb)
  Arms: Group A1 (hzVSF-v13 50mg, intravenous, single dose); Group A2 (hzVSF-v13 100mg, intravenous, single dose); Group A3 (hzVSF-v13 200mg, intravenous, single dose); Group A4 (hzVSF-v13 400mg, intravenous, single dose); Group A5 (hzVSF-v13 800mg, intravenous, single dose); Group A6 (hzVSF-v13 1200mg, intravenous, single dose)
Drug: hzVSF-v13 (subcutaneous, single dose) — Dosage form: 100mg of hzVSF-v13 (40 mg/mL in a 5 mL vial) Route: Subcutaneous Frequency: Dose at Day 1 (single administration)
  Other Names: a humanized monoclonal antibody (mAb)
  Arms: Group A7 (hzVSF-v13 100mg, subcutaneous, single dose)
Drug: hzVSF-v13 (intravenous, multiple dose) — Dosage form: 100mg / 400mg of hzVSF-v13 (40 mg/mL in a 5 mL vial) Route: Intravenous Frequency: Dose at Day 1, Day 15, Day 29, Day 43, Day 57 (multiple administration)
  Other Names: a humanized monoclonal antibody (mAb)
  Arms: Group B1 (hzVSF-v13 100mg, intravenous, multiple dose); Group B2 (hzVSF-v13 400mg, intravenous, multiple dose)
Drug: Placebo (intravenous, single dose) — Dosage form: 0.9% NaCl Solution Route: Intravenous Frequency: Dose at Day 1 (single administration)
  Other Names: 0.9% Normal saline
  Arms: Placebo (intravenous, single dose)
Drug: Placebo (subcutaneous, single dose) — Dosage form: 0.9% NaCl Solution Route: Subcutaneous Frequency: Dose at Day 1 (single administration)
  Other Names: 0.9% Normal saline
  Arms: Placebo (subcutaneous, single dose)
Drug: Placebo (intravenous, multiple dose) — Dosage form: 0.9% NaCl Solution Route: Intravenous Frequency: Dose at Day 1, Day 15, Day 29, Day 43, Day 57 (multiple administration)
  Other Names: 0.9% Normal saline
  Arms: Placebo (intravenous, multiple dose)

SUMMARY:
Assessment of the safety, tolerability and pharmacokinetics (PK) characterization of hzVSF-v13 with single and multiple doses (intravenous and subcutaneous) compared to placebo in healthy subjects.

DETAILED DESCRIPTION:
A phase I, double-blind, placebo-controlled, single and multiple dose

ELIGIBILITY:
Inclusion Criteria:

* Males or females (of either childbearing or non-childbearing potential), of any race, between 18 and 60 years of age, inclusive on day of screening.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive on day of screening.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline QTc interval at each time point | Group A1~A7: Day 1 (pre-dose), Day 8, Day 15, Day 22, Day 29, Day 36, Day 50, Day 64, Day 78, Day 92 Group B1~B2: Day 1 (pre-dose), Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 98, Day 162
  Safety assessments of hzVSF-v13 by ECG parameter (QTc interval), ECG Bandwidth: 100~300Hz

SECONDARY OUTCOMES:
Pharmacokinetic - Cmax | Group A1~A7: Predose, 0.25 ~ 2184 hours postdose Group B1~B2: Day 1 (predose ~ 48 hours postdose), Day8, Day15, Day29, Day43, Day 57 (predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 12, 24 hours postdose), Day71, Day85, Day98
  Maximum observed Concentration of hzVSF-v13
Pharmacokinetic - AUC0-∞ | Group A1~A7: Predose, 0.25 ~ 2184 hours postdose Group B1~B2: Day 1 (predose ~ 48 hours postdose), Day8, Day15, Day29, Day43, Day 57 (predose, 0.25, 0.5, 1, 2, 4, 6, 8, 10, 12, 24 hours postdose), Day71, Day85, Day98
  Area under the plasma concentration-time curve (AUC) from time zero to infinity

CONTACTS AND LOCATIONS:
Overall Officials: +61-8-70887900 Wabnitz, phD, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX, Clinical Research Pty Ltd., Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No